CLINICAL TRIAL: NCT00548769
Title: An Open-label, Randomised, Four Period Crossover Study to Investigate the Relative Pharmacokinetic Profiles of Tablets From Three Batches of Firategrast With Different Surface Areas and Two Different Tablet Formulations Containing the Same Batch of Firategrast, Given as Single 900mg Doses to Male and Female Subjects With a Diagnosis of Multiple Sclerosis
Brief Title: Firategrast (SB683699) Surface Area Study in Multiple Sclerosis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A4M109079
Record Dates: First submitted 2007-10-23; First posted 2007-10-24 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Multiple Sclerosis
Keywords: PK,; SB-683699,; multiple sclerosis; firategrast,; surface area,
MeSH Terms: conditions — Multiple Sclerosis | interventions — Firategrast; D-Worm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence ADBC (Experimental): Subjects will be administered formulation A, formulation D, formulation B and formulation C across four study days each separated by a washout period of at least seven days. Subjects will fast overnight prior to dosing. Blood samples will be collected at intervals over a period of 24 hours post-dose.
  Interventions: Drug: Formulation A; Drug: Formulation B; Drug: Formulation C; Drug: Formulation D
- Sequence BACD (Experimental): Subjects will be administered formulation B, formulation A, formulation C and formulation D across four study days each separated by a washout period of at least seven days. Subjects will fast overnight prior to dosing. Blood samples will be collected at intervals over a period of 24 hours post-dose.
  Interventions: Drug: Formulation A; Drug: Formulation B; Drug: Formulation C; Drug: Formulation D
- Sequence CBDA (Experimental): Subjects will be administered formulation C, formulation B, formulation D and formulation A across four study days each separated by a washout period of at least seven days. Subjects will fast overnight prior to dosing. Blood samples will be collected at intervals over a period of 24 hours post-dose.
  Interventions: Drug: Formulation A; Drug: Formulation B; Drug: Formulation C; Drug: Formulation D
- Sequence DCAB (Experimental): Subjects will be administered formulation D, formulation C, formulation A and formulation B across four study days each separated by a washout period of at least seven days. Subjects will fast overnight prior to dosing. Blood samples will be collected at intervals over a period of 24 hours post-dose.
  Interventions: Drug: Formulation A; Drug: Formulation B; Drug: Formulation C; Drug: Formulation D

INTERVENTIONS:
Drug: Formulation A — Formulation A will contain firategrast drug substance from native drug batch Irvine. Subjects will be administered three tablets of 300 milligrams with drug substance surface area of 2.1 square meter per gram. The tablets will be administered with 240 milliliters of water.
  Other Names: firategrast (SB683699)
Drug: Formulation B — Formulation B will contain firategrast drug substance from native drug batch Tonbridge. Subjects will be administered three tablets of 300 milligrams with drug substance surface area of 2.6 square meter per gram. The tablets will be administered with 240 milliliters of water.
Drug: Formulation C — Formulation C will contain firategrast drug substance from Tonbridge single pass micronized drug. Subjects will be administered three tablets of 300 milligrams with drug substance surface area of 3-4 square meter per gram. The tablets will be administered with 240 milliliters of water.
Drug: Formulation D — Formulation D will contain firategrast drug substance from Tonbridge with reduced tablet size. Subjects will be administered three tablets of 300 milligrams with drug substance surface area of 2.6 square meter per gram. The tablets will be administered with 240 milliliters of water.

SUMMARY:
Sufficient subjects with a confirmed diagnosis of MS (EDSS score of 6.5 or below), will be recruited to ensure that 30 subjects (approx. equal numbers of each gender) complete the study. Subjects will undergo a screening visit, then four study days, each separated by a washout period of at least 7 days, when the different firategrast batches of drug substance will be administered, and a follow-up visit.

DETAILED DESCRIPTION:
An open-label, randomised, four period crossover study to investigate the relative pharmacokinetic profiles of tablets from three batches of firategrast with different surface areas and two different tablet formulations containing the same batch of firategrast, given as single 900mg doses to male and female subjects with a diagnosis of Multiple Sclerosis

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18-65 years inclusive with a diagnosis of MS
* EDSS between 0-6.5 inclusive at the Screening visit
* QTc <450msec
* A female subject is eligible to enter the study if she is of non-childbearing potential, or of childbearing potential, has a negative urine pregnancy test at Screening, and agrees to consistent and correct use of adequate contraception
* Provide a signed and dated written informed consent prior to study participation
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions
* A negative urine drugs of abuse test.
* No evidence of pulmonary tuberculosis as verified by a negative chest X-ray within the past 6 months

Exclusion Criteria:

* Subjects receiving corticosteroids within 4 weeks of Screening for treatment of MS. If non-systemic steroids are being used for other chronic inflammatory conditions, subjects may be included at the discretion of the investigator after discussion with the GSK medical monitor.
* Use of an β-interferon product, glatiramer acetate or azathioprine within 3 months of Screening, or use of Mitoxantrone within 12 months of Screening. Subjects who have received other therapies affecting the immune system (such as IVIg, cyclophosphamide, plasmapheresis, or any other immunosuppressive or immunomodulatory treatment) in the past may be included on a case by case basis after discussion with the GSK medical monitor. None of these treatments will be allowed during this study
* Previous exposure to alemtuzumab, natalizumab or bone marrow transplantation or whole body irradiation.
* Subjects with a cardiac pacemaker or any other type of metal implant or with any other contraindication for MRI (including known allergy to gadolinium).
* Use of 4-aminopyridine, rosiglitazone, pioglitazone and any other compounds metabolised primarily through cytochrome P450 2C8 are prohibited at Screening and throughout the study
* Subjects with clinically significant renal laboratory values: subjects with a calculated creatinine clearance <60ml/min
* Subjects with local urinalysis findings outside of ranges defined in the protocol during the screening period.
* Presence of clinically significant hepatic laboratory values
* CD4 count <500 cells/µl, CD4:CD8 <1.0, idiopathic CD4/CD8 lymphopenia or secondary lymphopenia at Screening.
* JCV DNA detected in plasma or buffy coat using PCR
* Any findings on the MRI of the brain other than MS, except for benign findings that require no further evaluation or treatment and do not have an impact on the patient's neurological health
* Current or history of cancer, excluding localized non-melanoma skin cancer.
* Uncontrolled or any active bacterial, viral, or fungal infection. Any previous serious infections should be discussed with the GSK medical monitor (e.g. opportunistic or atypical infections).
* History of tuberculosis or positive chest X-ray for TB
* Known congenital or acquired immunodeficiency.
* Any abnormality on 12-lead ECG at Screening which is clinically significant in the opinion of the investigator.
* Subjects with positive hepatitis B, hepatitis C or HIV tests at Screening.
* Women who are lactating, pregnant (positive pregnancy test at Screening), or planning to become pregnant during the course of the study.
* Recent history or suspicion of current drug abuse (including analgesic abuse) or alcohol abuse within the last 6 months prior to Screening.
* Use of an investigational drug for condition other than MS within 30 days or 5 half-lives (whichever is longer) preceding Screening. Prior use of an investigational drug for MS should be discussed with the GSK medical monitor.
* Any concurrent illness, disability or clinically significant abnormality (including laboratory tests) that may affect the interpretation of clinical efficacy or safety data or prevent the subject from safely completing the assessments required by the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-04-21 (Actual); Primary Completion 2007-11-26 (Actual); Study Completion 2007-11-26 (Actual)

PRIMARY OUTCOMES:
The AUC(0-24) for firategrast following administration of tablets made from three different batches of drug with different surface areas. | Pre-dose. 0.5 hours, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 16 hours, 24 hours post dose

SECONDARY OUTCOMES:
Cmax and Tmax. The AUC(0-24) Cmax and Tmax of of SB683699 metabolite GW786375X. | Pre-dose. 0.5 hours, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 16 hours, 24 hours post dose
AEs, vital signs and clinical laboratory data during the course of the study. | Throughout the course of the study
SB-683699 and GW786375X plasma concentration to derive pharmacokinetic parameters. | Pre-dose. 0.5 hours, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 16 hours, 24 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- GSK Investigational Site, Prague, Czechia
- GSK Investigational Site, Berlin, Germany
- Poland (2):
  - GSK Investigational Site, Grodzisk Mazowiecki
  - GSK Investigational Site, Poznan

REFERENCES:
- See also: Results for study 109079 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/A4M109079?search=study&search_terms=A4M109079#rs